CLINICAL TRIAL: NCT03471767
Title: A Randomized, Double-Blind 4-Week Study to Evaluate the Impact of AXS-05 on Smoking Behavior
Brief Title: AXS-05 Phase II Trial on Smoking Behavior
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James Davis (Other)
Collaborators: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, James Davis, Medical Director, Duke Center for Smoking Cessation, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00089413
Record Dates: First submitted 2018-03-19; First posted 2018-03-21 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Smoking Cessation; Smoking, Cigarette; Nicotine Dependence
Keywords: Smoking cessation; Nicotine dependence; Bupropion; DXM; Nicotine addiction; Cigarette smoking; Dextromethorphan
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking; Tobacco Use Disorder | interventions — Bupropion; Dextromethorphan

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either take AXS-05 or BUP SR in parallel for the duration of the study.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AXS-05 (Experimental): Participants will receive AXS-05 (Dextromethorphan Immediate Release + Bupropion Sustained Release) for 4 weeks and will be instructed to take 1 tablet two times per day, at least 8 hours apart and 1 hour prior to a meal, and 2 hours after a meal.
  Interventions: Drug: AXS-05
- Bupropion SR (Active Comparator): Participants will receive Bupropion SR (Bupropion Sustained Release) for 4 weeks and will be instructed to take 1 tablet two times per day, at least 8 hours apart and 1 hour prior to a meal, and 2 hours after a meal.
  Interventions: Drug: Bupropion SR

INTERVENTIONS:
Drug: AXS-05 — Dextromethorphan Immediate Release + Bupropion Sustained Release: Take 1 tablet two times per day, at least 8 hours apart and 1 hour prior to a meal, and 2 hours after a meal.
  Other Names: Bupropion/dextromethorphan
  Arms: AXS-05
Drug: Bupropion SR — Bupropion Sustained Release: Take 1 tablet two times per day, at least 8 hours apart and 1 hour prior to a meal, and 2 hours after a meal.
  Other Names: Wellbutrin SR; Zyban SR
  Arms: Bupropion SR

SUMMARY:
This research study is designed with the purpose of evaluating a new drug, combination Dextromethorphan-Bupropion (AXS-05), for its effects on smoking behavior.

DETAILED DESCRIPTION:
This study aims to investigate the potential efficacy of a combination of two FDA-approved agents, sustained release (SR) Bupropion (BUP) and immediate release (IR) Dextromethorphan (DXM), for the purpose of smoking cessation treatment. DXM, a widely used over-the-counter cough suppressant, is a nicotine receptor antagonist. In fact, studies by Duke's Center for Smoking Cessation (CSC) have shown that administration of DXM leads to a decrease in self-administration of nicotine in nicotine-dependent rats. DXM, however, has not been studied in humans. DXM, when taken alone, is not expected to be useful for treating nicotine dependence in humans given DXM rapidly metabolizes in humans via CYP2D6. As a result, therapeutic concentrations needed to bind to nicotine receptors are not obtained. Therapeutic concentrations of DXM are required, therefore, to allow DXM to bind to nicotine receptors and act as a nicotine antagonist. In order to attain therapeutic concentrations of DXM a metabolism inhibitor must be introduced. BUP is a well-known FDA approved smoking cessation medication that has been shown to inhibit the metabolism of DXM. When BUP is co-administered with DXM to healthy volunteers, a significant increase in DXM plasma levels is observed.

Currently, Axsome Therapeutics Inc. (Axsome) is developing and testing an oral fixed-dose combination of IR DXM with SR BUP to achieve therapeutic concentrations of DXM. This investigational drug has been named AXS-05. Axsome has found AXS-05 to be generally safe and well-tolerated in three Phase 1 studies. The adverse event profile of AXS-05 was similar to that of BUP alone.

Given the distinct mechanisms by which BUP and DXM interact, it is hoped that combining DXM and BUP will prove more efficacious than either drug administered alone for the purpose of tobacco use treatment in humans.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 18 years or above
2. Daily smoker using 10 or more cigarettes per day
3. Willing to be smoke-free for 7 days
4. Is able to provide written informed consent (in English) to participate in the study and able to understand the procedures and study requirements.
5. Is willing to voluntarily sign and date an informed consent form that is approved by an institutional review board before the conduct of any study procedure.

Key Exclusion Criteria:

1. Current use of a smoking cessation medication (e.g. nicotine replacement, Varenicline, bupropion)
2. Current use of tobacco product other than cigarettes (e.g. e-cigarettes, smokeless tobacco)
3. Not pregnant or breastfeeding
4. Contraindication to the use of bupropion.
5. Additional criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Davis, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke Center for Smoking Cessation, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AXS-05: AXS-05: Dextromethorphan Immediate Release + Bupropion Sustained Release: Take 1 tablet two times per day, at least 8 hours apart and 1 hour prior to a meal, and 2 hours after a meal for 4 weeks.
- Bupropion SR: Bupropion SR: Bupropion Sustained Release: Take 1 tablet two times per day, at least 8 hours apart and 1 hour prior to a meal, and 2 hours after a meal for 4 weeks
Period: Overall Study
Arm/Group | AXS-05 | Bupropion SR
Started | 31 | 27
Completed | 25 | 23
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — PI Withdrawal | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AXS-05 | Bupropion SR | Total
Number analyzed (Participants) | 31 | 27 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.03 (13.61) | 46.48 (11.34) | 48.38 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 15 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 30 | 25 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 15 | 23
  White | 22 | 11 | 33
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 27 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in Smoking Intensity
Description: Smoking intensity refers to the number of cigarettes smoked per day.
Time Frame: Baseline (V1), 3-Week Follow-Up Visit (V4)
Measure: Mean (Standard Error); unit: change in cigarettes per day
Arm/Group | AXS-05 | Bupropion SR
Number analyzed (Participants) | 31 | 27
change in cigarettes per day | -8.49 (0.37) | -6.79 (0.39)
Statistical Analysis 1: Comparison: AXS-05 vs Bupropion SR; Test type: Superiority — Multilevel modeling (MLM) was used to model daily reports of cigarettes smoked as a function of week, treatment (AXS-05 vs. bupropion), and the interaction between week and treatment. The contrast between the two treatment groups in change in smoking intensity from baseline to week 3 was estimated within the context of the model; p = 0.05, t-test, 2 sided — This was not adjusted for multiple comparisons, because the primary hypothesis was established a-priori; Mean Difference (Final Values) = -1.70, 95% CI 2-sided [-2.75 to -0.65], Standard Error of Mean 0.54

2. Secondary Outcome: Change in Smoking Behavior
Description: 7-day point prevalence smoking abstinence. Measured by composite self-report diaries and biochemically confirmed via expired CO and salivary cotinine.
Time Frame: 3-Week Follow-Up Visit (V4), 4-Week Follow-Up Visit (V5)
Population: Not all participants participated in this abstinence test.
Measure: Count of Participants; unit: Participants
Arm/Group | AXS-05 | Bupropion SR
Number analyzed (Participants) | 24 | 18
Participants | 16 | 12

3. Secondary Outcome: Medication Adherence
Description: Medication adherence is measured by composite self-reported diaries.
Time Frame: Baseline (V1), 3-Week Follow-Up Visit (V4)
Population: Not all participants participated in the full reporting period (dropped out or withdrew).
Measure: Mean (Standard Deviation); unit: percentage of adherence
Arm/Group | AXS-05 | Bupropion SR
Number analyzed (Participants) | 30 | 23
percentage of adherence | 97.08 (5.97) | 96.60 (5.27)

4. Secondary Outcome: Medication Tolerance by Self-Reported Side Effects
Description: Number of participants who scored 3 or higher on a 7-point Likert scale ranking severity of side effects (1-2 mild; 3-5 moderate; 6-7 severe).
Time Frame: Baseline (V1), 3-Week Follow-Up Visit (V4)
Measure: Count of Participants; unit: Participants
Arm/Group | AXS-05 | Bupropion SR
Number analyzed (Participants) | 31 | 27
Participants | 7 | 5

5. Secondary Outcome: Medication Tolerance by Serious Adverse Events
Description: Measured by FDA reporting guidelines on adverse event or serious adverse event designation.
Time Frame: Baseline (V1), 4-Week Follow-Up Visit (V5)
Population: There were no study-related serious adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | AXS-05 | Bupropion SR
Number analyzed (Participants) | 31 | 27
Participants | 0 | 0

6. Secondary Outcome: Urinary Levels of Dextromethorphan
Description: Measured via Urinary Dextromethorphan testing.
Time Frame: 3-Week Follow-Up Visit (V4)
Population: Data not collected on the Bupropion SR group. Some individuals in the AXS-05 group had missing data or withdrew/dropped out early.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AXS-05 | Bupropion SR
Number analyzed (Participants) | 29 | 0
ng/mL | 1902.1 (1304.4) |

7. Primary Outcome: Percentage of Participants Who Experienced a More Than 50% Reduction in Expired Carbon Monoxide (CO) Levels
Description: A biochemical marker of smoking intensity.
Time Frame: Baseline (V1), 3-Week Follow-Up Visit (V4)
Measure: Number; unit: percentage of participants
Arm/Group | AXS-05 | Bupropion SR
Number analyzed (Participants) | 31 | 27
percentage of participants | 52.0 | 30.4
Statistical Analysis 1: Comparison: AXS-05 vs Bupropion SR; Test type: Other; p = 0.15, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Approximately four weeks
Arm/Group | AXS-05 | Bupropion SR
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/31 | 1/27
Other Adverse Events (participants affected / at risk) | 4/31 | 8/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-05 (N=31) | Bupropion SR (N=27)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) — Non-study related; no show to final study visit, contact attempts unsuccessful. Approximately 1 month post-stroke, contact made. Verbal consent given to review medical chart. Deemed not study related.
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) — Hospitalized for urinary tract infection. Past history of UTI's. Deemed not study related.
Broken Jaw (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Fell down stairs and sustained broken jaw. Deemed not study related.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AXS-05 (N=31) | Bupropion SR (N=27)
Dry Mouth (Gastrointestinal disorders) | 2 | 3
Headache (Nervous system disorders) | 0 | 2
Insomnia/Sleep Disturbance (Psychiatric disorders) | 2 | 2
Abnormal/Vivid Dreams (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT03471767/Prot_SAP_000.pdf